CLINICAL TRIAL: NCT05217082
Title: Health-Related Quality of Life (HRQoL) in Patients With Relapsed and/or Refractory Multiple Myeloma (RRMM) With Triple Class Exposure in Japan
Brief Title: A Study Assessing the Health-Related Quality of Life (HRQoL) in Participants With Relapsed and/or Refractory Multiple Myeloma (RRMM) With Triple Class Exposure
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA089-013
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; HRQoL; Relapsed; Refractory; Outcomes
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with relapsed/refractory multiple myeloma (RRMM) who have already received a proteasome inhibitor, an immunomodulatory agent, and an anti-CD38 antibody

SUMMARY:
The purpose of this observational study is to assess HRQoL in relapsed and/or refractory multiple myeloma (RRMM) participants who have previously received a proteasome inhibitor, an immunomodulatory agent, and an anti-CD38 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Must have sufficient command of the Japanese language to understand the study instructions and requirements
* Must be a resident of Japan
* Must have received prior treatment with:

  1. a proteasome inhibitor,
  2. an immunomodulatory agent, and
  3. an anti-CD38 antibody Subjects must be either 2-4 months, 5-7 months, or 8-11 months post triple class therapy exposure at time of consent
* Subject must be diagnosed with multiple myeloma

Exclusion Criteria:

* Participants enrolled in a clinical trial that includes at least one novel/ experimental agent at the point of questionnaire completion

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will consist of approximately 50 participants diagnosed with relapsed/refractory multiple myeloma (RRMM) with triple class therapy exposure identified by physicians.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQoL) in specific domains: Fatigue, as measured by EORTC QLQ-C30 | Up to 1 year
  EORTC QLQ-C30 defined as European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30
HRQoL in specific domains: Pain, as measured by the EORTC QLQ-C30 | Up to 1 year
HRQoL in specific domains: Physical Functioning as measured by the EORTC QLQ-C30 | Up to 1 year
HRQoL in specific domains: Cognitive Functioning, as measured by the EORTC QLQ-C30 | Up to 1 year
HRQoL in specific domains: Global health, as measured by the EORTC QLQ-C30 | Up to 1 year
HRQoL in specific domains: Disease Symptoms as measured by the EORTC QLQ-MY20 | Up to 1 year
  EORTC QLQ-MY20 defined as European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-MY20
HRQoL in specific domains: Side effects as measured by the EORTC QLQ-MY20 | Up to 1 year

SECONDARY OUTCOMES:
HRQoL in specific domains: Functional Scale as measured by the EORTC QLQ-C30 | Up to 1 year
HRQoL in specific domains: Symptoms Scale as measured by the EORTC QLQ-C30 | Up to 1 year
HRQoL in specific domains: Global Health Status as measured by the EORTC QLQ-C30 | Up to 1 year
HRQoL in specific domains: Future Perspective as measured by the EORTC QLQ-MY20 | Up to 1 year
HRQoL in specific domains: Body Image as measured by the EORTC QLQ-MY20 | Up to 1 year
HRQoL in specific domains: Generic HRQoL as measured by the EQ-5D-5L | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Morrisville, North Carolina, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome